CLINICAL TRIAL: NCT05291338
Title: Pharmacogenetic Study in Hepatocellular Carcinoma Patients Underwent TACE
Brief Title: Pharmacogenetic Study in Hepatocellular Carcinoma Patients.
Status: Completed | Type: Observational
Sponsor: Rehab Werida (Other)
Responsible Party: Sponsor-Investigator, Rehab Werida, Principal Investigator, Damanhour University
Organization: Damanhour University (Other)
Other Study IDs: genetic in hepatic cancer
Record Dates: First submitted 2022-03-12; First posted 2022-03-22 (Actual); Last update posted 2023-07-28 (Actual); Status verified 2023-07

CONDITIONS: Hepatocellular Carcinoma
Keywords: ANG-2; IL28B; genetic polymorphisms
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Doxorubicin; Ethiodized Oil

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- HCC patients: 116 hepatocellular carcinoma patients underwent TACE
  Interventions: Drug: Doxorubicin; Drug: Lipiodol

INTERVENTIONS:
Drug: Doxorubicin — no optimal dosage of doxorubicin in TACE procedures (ranging from 30 to 75 mg/m2 up to a maximum of 150 mg/m2 ) according to tumor size
  Other Names: Adriamycin
Drug: Lipiodol — Lipiodol dose should be over 5 ml if tumor diameter is less than 5 cm, and the maximum dose will be 10 ml when the tumor develops to more than 5 cm in diameter.
  Other Names: ethiodized oil

SUMMARY:
evaluate the prognostic value of genetic polymorphisms in HCC Egyptian patients undergoing TACE using lipiodol and doxorubicin.

DETAILED DESCRIPTION:
Research Objectives This study aims to determine the predictive effect of ANG-2 and IL28B genetic polymorphisms in safety and efficacy of doxorubicin and lipiodol used for the treatment of Egyptian HCC patients. Moreover, this study will determine the association between genetic polymorphisms of ANG-2 and IL28B with HCC severity.

Patients & Methods Study design Our study is a prospective study for HCC patients undergoing TACE of doxorubicin and lipiodol.

Sample Size Based on previous published incidence of gene it will be at least 116 patients. Efficacy and Safety

1. Target lesions response will be measured according to modified Response Evaluation Criteria in Solid Tumors (RECIST) to (15):

   Complete response, Partial response, Progressive disease and Stable disease.
2. Repeated TACE sessions will be planned individually based on the tumor response to the treatment protocol.
3. Follow up will be performed for detection of tumor size using triphasic CT scan as a measure of efficacy. Moreover, all patients will be reevaluated for CBC, liver and kidney functions, in the follow up visit, to detect incidence of any adverse effects.
4. Patients will be asked for any side effects such as (myelosuppression, anorexia, nausea, vomiting, and/or alopecia).
5. Patients will be followed for progression-free survival after receiving TACE.

Method & Proposal Steps

1. Approval will be obtained from Research Ethics Committee of Faculty of Pharmacy, Damanhour University.
2. Patients will be recruited from Ain Shams University hepatoma group, EL Demerdash Hospital, Cairo, Egypt.
3. At baseline and follow up visits after TACE, all patients will be assessed for complete blood count (CBC), kidney function, liver function, liver enzymes, alpha fetoprotein (AFP) and viral markers. Moreover, triphasic pelviabdominal CT will be performed before and after TACE.
4. Serum samples will be collected for ANG-2 and IL28B genotyping.
5. Genetic polymorphisms of ANG-2 and IL28B will be detected by real time polymerase chain reaction (RT-PCR).

   * Five mls of whole blood will be collected then separation of plasma will be performed.
   * Extraction of genomic DNA from blood samples by DNA extraction kit.
   * DNA qualification will be performed by Nano drop.
   * Genotyping will be done by allelic discrimination using Taqman assays specific for each polymorphism.
   * Assays will be done according to manufacturer protocol using real time PCR machine.
6. All patients will receive lipiodol and doxorubicin during TACE. Doxorubicin dose will differ among patients according to tumor size, patient condition, patient's laboratory data and presence of hepatic arteriovenous fistula.
7. Appropriate statistical tests will be conducted to evaluate the significance of the results.
8. Results, conclusion, discussion and recommendations will be given.

ELIGIBILITY:
Inclusion Criteria:

* Eligible patients should fulfill the following criteria:

  1. A diagnosed HCC patient.
  2. Age ≥20 years.
  3. Patients with adequate organ function.
  4. HCC not eligible for curative measures (radiofrequency, microwave and surgery).

Exclusion Criteria:

* Patient will be excluded for any of the following:

  1. Patients refused to sign the written consent.
  2. Age > 75 years.
  3. The presence of major portal vein thrombosis.
  4. Extrahepatic metastases.
  5. Hepatic encephalopathy.
  6. Current infection.
  7. Gastrointestinal bleeding within a month.
  8. Uncontrolled ascites.
  9. Serum bilirubin > 3.0 mg/dl, serum albumin < 2.8 g/dl, serum creatinine concentration > 1.5 mg/dl, white blood cell counts < 3,000/mm3 and platelet counts < 30,000/mm3.
  10. Patients with other types of malignancy, advanced organ failure, and advanced medical co-morbidity.
  11. Pregnant females.

Ages: 20 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Egyptian HCC patients on doxorubicin and lipiodol treatment
Sampling Method: Probability Sample
Enrollment: 107 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-04-01 (Actual)

PRIMARY OUTCOMES:
Angiopoietin (ANG-2) rs55633437. | 1 month
  Gene
Interleukin 28 B (IL28B) rs12979860. | 1 month
  Gene

CONTACTS AND LOCATIONS:
Overall Officials: Rehab H Werida, Ass Prof., Study Director — Damanhour University
Locations (1):
- Ain Shams University hepatoma group, EL Demerdash Hospital, Cairo, Egypt., Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Marisi G, Petracci E, Raimondi F, Faloppi L, Foschi FG, Lauletta G, Iavarone M, Canale M, Valgiusti M, Neri LM, Ulivi P, Orsi G, Rovesti G, Vukotic R, Conti F, Cucchetti A, Ercolani G, Andrikou K, Cascinu S, Scartozzi M, Casadei-Gardini A. ANGPT2 and NOS3 Polymorphisms and Clinical Outcome in Advanced Hepatocellular Carcinoma Patients Receiving Sorafenib. Cancers (Basel). 2019 Jul 20;11(7):1023. doi: 10.3390/cancers11071023. PMID 31330833
- [Background] Rashed WM, Kandeil MAM, Mahmoud MO, Ezzat S. Hepatocellular Carcinoma (HCC) in Egypt: A comprehensive overview. J Egypt Natl Canc Inst. 2020 Jan 16;32(1):5. doi: 10.1186/s43046-020-0016-x. PMID 32372179
- [Derived] Werida RH, Abd El Baset OA, Askar S, El-Mohamdy M, Omran GA, Hagag RS. Efficacy of doxorubicin and lipiodol therapy by trans-arterial chemoembolization in hepatocellular carcinoma Egyptian patients and relation to genetic polymorphisms. Expert Rev Anticancer Ther. 2024 Oct;24(10):1009-1020. doi: 10.1080/14737140.2024.2391364. Epub 2024 Aug 21. PMID 39138591